CLINICAL TRIAL: NCT07276880
Title: Preoperative Chemotherapy, Pembrolizumab and Low or High Dose RADiation in an Expansion Cohort of Node(+), Triple Negative Breast Cancer
Acronym: P-RAD(+)TN-DCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2426-DCT; R01CA274254 (NIH)
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer (TNBC); HER2-Negative Breast Carcinoma; Node-positive Breast Cancer
Keywords: radiation therapy; neoadjuvant treatment; pembrolizumab; immune checkpoint inhibitor; radiotherapy boost
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: hybrid decentralized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM 1 (Experimental): Participants will receive a low dose radiation therapy boost in 3 fractions (3Gy x 3 fraction = 9Gy total).
  Interventions: Drug: Neoadjuvant Pembrolizumab; Radiation: low dose neoadjuvant boost
- ARM 2 (Experimental): Participants will receive a high dose radiation therapy boost in 3 fractions (8Gy x 3 fraction = 24Gy total).
  Interventions: Drug: Neoadjuvant Pembrolizumab; Radiation: High dose neoadjuvant boost

INTERVENTIONS:
Drug: Neoadjuvant Pembrolizumab — 200 milligrams per square meter Neoadjuvant Pembrolizumab will be administered intravenously.
Radiation: low dose neoadjuvant boost — An external beam radiotherapy boost of 9Gy total will be administered over 3 fractions.
  Arms: ARM 1
Radiation: High dose neoadjuvant boost — An external beam radiotherapy boost of 24Gy total will be administered over 3 fractions.
  Arms: ARM 2

SUMMARY:
This is a prospective radiation dose-finding, phase 2 expansion study of the Triple Negative (TN) cohort of the multicenter randomized study P-RAD (A Randomized Study of Preoperative Chemotherapy, Pembrolizumab and No, Low or High Dose RADiation in Node-Positive, HER2-Negative Breast Cancer; NCT04443348) that seeks to establish the optimal dose of radiation therapy (RT) to elicit an immune response when combined with immune checkpoint inhibitor (ICI) in breast cancer patients. Eligible subjects include women or men with operable, lymph node-positive, triple negative (TN) breast cancer who are candidates for standard of care neoadjuvant chemo-immunotherapy (NAC) based on the KEYNOTE-522 clinical trial. Thirty-two (n=32) patients will be randomized 1:1 to receive either low RT boost (9Gy total) or high RT boost (24Gy total). All RT will be delivered to the intact breast tumor in 3 daily fractions over 3 days.

In the Neoadjuvant Phase, the first cycle (C1) of pembrolizumab (200 mg i.v.) will be administered within 0-2 days of initiating RT. Participation in this study requires availability of residual diagnostic tissue biopsies of the primary tumor and metastatic lymph node for research use. If this tissue is not available, baseline research biopsies will be performed. Additionally, a research biopsy of the breast tumor and lymph node is required on Day 10-14 of C1 of pembrolizumab. After completion of the research biopsy in Week 2, the participants can commence standard-of-care neoadjuvant chemotherapy and pembrolizumab at the discretion of their medical oncology provider. After completing NAC, participants will undergo standard of care surgical resection of the breast and axillary lymph nodes, at the discretion of their surgical oncology provider. In the Adjuvant Phase, participants will receive standard of care adjuvant systemic therapy and standard of care adjuvant radiotherapy (if indicated), although recognizing that the breast tumor boost portion of this treatment has already been administered preoperatively. Except for late radiation adverse reactions of special interest, which will be followed yearly for up to 5 years, follow-up will occur every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a subject must meet all of the eligibility criteria outlined below.

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information. Subjects are willing and able
* to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at the time of consent.
* ECOG or Karnofsky Performance Status of 0 or 1

Exclusion Criteria:

* Active infection requiring systemic therapy.
* Pregnant or breastfeeding.
* Prior ipsilateral invasive breast, chest wall or thoracic radiotherapy
* Prior ipsilateral invasive breast cancer, contralateral breast cancer or a known
* additional, invasive malignancy that is progressing or required active treatment in
* the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Nodal Pathologic Complete Response rate(pCR) | Time of surgery (24 week)
  Nodal pCR is defined in a patient with no residual cancer cells in all sampled regional lymph nodes following completion of neoadjuvant systemic therapy as assessed by the study pathologist at the time of definitive surgery.
  Nodal pCR rates will be calculated and analyzed separately for patients receiving low versus high dose RT. A pooled analysis, incorporating the corresponding (3Gyx3 or 8Gyx3) patient cohort from the P-RAD trial, will be performed.

SECONDARY OUTCOMES:
The CD3+/CD8+ T cell Breast post-treatment biopsy | Time of surgery (24 week)
  The CD3+/CD8+ T cell Breast Immunoscore of post-treatment biopsy samples represents an average of percentage ranked scores for (i) CD3+ density in intra-tumoral region, (ii) CD3+ density in peri-tumoral region, (iii) CD8+ density in intra-tumoral region, and (iv) CD8+ density in peri-tumoral region. The reference cohort for determining percentage ranks will be the pre-treatment biopsy samples.
Composite pathologic complete response (pCR) (ypT0/Tis ypN0) | Time of surgery (24 week)
  Composite pCR =T0/Tis and pN0 will be defined as the percentage of patients with Tis/T0 disease in the breast and no evidence of residual cancer cells in all sampled regional lymph nodes following completion of neoadjuvant systemic therapy, assessed by the study pathologist at the time of definitive surgery.
Total residual cancer burden (RCB) | Time of surgery (24 week)
  RCB will be evaluated by the study pathologist and defined based on residual tumor size and/or area, overall cellularity, and extent of lymph node involvement.
Nodal pathologic complete response (pCR) | Time of surgery (24 week)
  Nodal pCR is defined as absence of residual cancer cells in all sampled regional lymph nodes.
Composite pathologic complete response (pCR) | Time of surgery (24 week)
  Composite pCR rate is measured by ypTis/T0 disease in the breast and the absence of residual cancer cells in all sampled regional lymph nodes.
Changes in pre- versus post-treatment intra-tumoral, peri-tumoral, and stromal CD3+ or CD8+ T cell percentages | Time of surgery (24 week)
  Intra-tumoral, peri-tumoral, and stromal CD3+ and CD8+ T-cell densities will be measured in biopsy and surgical specimens and compared. Pan-cytokeratin staining will be used to identify tumor regions, and the percentages will be analyzed.
Change in tumor-infiltrating lymphocyte (TIL) | Time of surgery (24 week)
  Tumor-infiltrating lymphocyte (TIL) counts will be assessed on hematoxylin and eosin (H&E)-stained biopsy and surgical specimens using the Salgado criteria, which evaluate the percentage of stromal area occupied by lymphocytes following standardized guidelines. The values in biopsy and surgical specimens and compared.
Change in Programmed cell death 1 ligand 1(PD-L1) | Time of surgery (24 week)
  Changes in PD-L1 expression levels will be assessed using the U.S. FDA-approved 22C3 pharmDx companion diagnostic assay to determine the Combined Positive Score (CPS). A CPS greater than 1 will be considered PD-L1 positive. The values in biopsy and surgical specimens and compared.
Changes in intratumoral, peri-tumoral, and stromal CD4+Foxp3+ T regulatory cell densities | Time of surgery (24 week)
  Changes in intratumoral, peri-tumoral, and stromal CD4+FOXP3+ regulatory T-cell densities will be quantified using quantitative immunofluorescence (QIF) for CD4 and FOXP3 in formalin-fixed, paraffin-embedded (FFPE) tumor biopsy and surgical specimens. Pan-cytokeratin staining will be used to identify tumor regions.
Adverse Events | Up to 60 weeks
  Adverse events will be classified and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0), at 30 days after investigational pembrolizumab administration. The number of observed AEs will be reported.
Invasive disease-free survival (iDFS) | Up to 5 years
  iDFS will be defined as the time from completion of surgery to the first occurrence of the following events: invasive ipsilateral, local, regional, or distant recurrence, or death due to breast cancer.
Event-free survival (EFS) | Up to 5 years
  EFS will be defined as the time from the initiation of the study treatment to any of the following events: progression of disease (precluding surgery), recurrence (local or distant), or death due to any cause.
Quality of life Global Health PROMIS in Low Dose Radiotherapy Boost Group | Baseline, Week 2, Week 8, Week 14, and Week 20, 6 months post-surgery, and monthly for up to 3 years
  Quality of life will be assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) tool developed by the National Institutes of Health (NIH) before and after treatment. It is designed to measure a patient's overall physical, mental, and social health using a brief and standardized questionnaire. Responses are collected using a 5-point Likert scale (1 = Poor, 5 = Excellent), summed into raw scores, and converted to standardized T-scores (mean = 50, SD = 10; range ~20-80), with higher scores indicating better health.
Quality of life BREAST-Q in Low Dose Radiotherapy Boost Group | Baseline, Week 2, Week 8, Week 14, and Week 20, 6 months post-surgery, and monthly for up to 3 years
  Patient-reported outcomes related to breast surgery will be assessed using the BREAST-Q questionnaire, a validated instrument measuring satisfaction with breasts, psychosocial well-being, physical well-being, and sexual well-being. Most items are answered on a 4- to 5-point Likert scale, for example: Satisfaction: "Very dissatisfied" → "Very satisfied" or Frequency/impact: "Never" → "Always" or "Not at all" → "Very much. "Responses are scored according to the BREAST-Q scoring system and transformed to a 0-100 scale, with higher scores indicating greater satisfaction or better quality of life.
The Was It Worth It (WIWI) in Low Dose Radiotherapy Boost Group | Baseline, Week 2, Week 8, Week 14, and Week 20, 6 months post-surgery, and monthly for up to 3 years
  The Was It Worth It (WIWI) instrument, also called the Trial Satisfaction survey, is a validated patient-reported outcome measure designed to assess participants' experiences and satisfaction with clinical trial participation. It evaluates whether patients feel that joining the trial was worthwhile and captures their overall perception of the trial experience. Responses are collected using a Likert-type scale (3 to 5 points) or categorical options, with higher scores indicating a more positive perception of trial participation. Scores will be summarized to assess overall patient satisfaction and the perceived value of trial involvement.
Quality of life Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) in Low Dose Radiotherapy Boost Group | Baseline, Week 2, Week 8, Week 14, and Week 20, 6 months post-surgery, and monthly for up to 3 years
  PRO-CTCAE, which collects information on the frequency, severity, interference, and presence or absence of symptoms such as pain, fatigue, nausea, and cutaneous side effects including rash and hand-foot syndrome. These toxicities are selected because they can be meaningfully reported from the patient perspective. PRO-CTCAE responses are scored from 0 to 4, or 0/1 for absent/present items. If the first response in an item set is the lowest on the scale (e.g., 'Never' for frequency or 'None' for severity), any conditionally branched items are scored as 0 and not treated as missing.
Comparison tumor-infiltrating lymphocyte (TIL) | Time of surgery (24 week)
  Differences in tumor-infiltrating lymphocyte (TIL) between low and high dose levels will be assessed by hematoxylin and eosin (H&E)-stained biopsy and surgical specimens using the Salgado criteria, which evaluate the percentage of stromal area occupied by lymphocytes following standardized guidelines. The values in biopsy and surgical specimens and compared. Differences in TIL between low and high dose levels (3Gyx3 or 8Gyx3) will be assessed by H&E.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Casey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials